CLINICAL TRIAL: NCT02344368
Title: The Effect of Sucrose on Pain Relief During Venous Blood Sampling in Preterm Infants: a Comparison of Two Different Doses
Brief Title: The Effect of Sucrose on Pain Relief During Venous Blood Sampling in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Lower Umfolozi Regional War Memorial Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/2089
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2016-07

CONDITIONS: Pain
Keywords: Sucrose; Anesthesia; Blood specimen collection; Injections, Intravenous
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.2 ml sucrose (Experimental): on 2 occasions within 1 week 0.2 ml sucrose 25% or 0.5 ml sucrose 25% will be given in randomized order to the same infant during blood sampling
  Interventions: Other: 0.2 ml sucrose 25%; Other: 0.5 ml sucrose 25%
- 0.5 ml sucrose (Experimental): on 2 occasions within 1 week 0.2 ml sucrose 25% or 0.5 ml sucrose 25% will be given in randomized order to the same infant during blood sampling
  Interventions: Other: 0.2 ml sucrose 25%; Other: 0.5 ml sucrose 25%

INTERVENTIONS:
Other: 0.2 ml sucrose 25% — Administered on the tongue by a syringe, a half dose two minutes before blood sampling and the other half dose immediately before sampling
Other: 0.5 ml sucrose 25% — Administered on the tongue by a syringe, a half dose two minutes before blood sampling and the other half dose immediately before sampling

SUMMARY:
Despite the fact that oral sucrose is the most frequently studied non-pharmacological intervention for procedural pain relief in infants, there is a paucity of data on the minimal effective dose. The aim of this study is to find the minimal effective dose of sucrose to reduce pain during a single venous blood sampling procedure.

ELIGIBILITY:
Inclusion Criteria:

* born preterm
* more than 1000 gram

Exclusion Criteria:

* severe intraventricular hemorrhage
* cerebral malformations
* other malformations requiring surgery
* medication that may impair pain expression (opioids, paracetamol, sedatives)

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
pain | 1 week
  assessed by Premature Infant Pain Profile-Revised (PIPP-R). Pain score related to the blood sampling will be performed two times: at skin puncture and immediately after the needle has been removed

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Bergseng, MD PhD, Study Director — Norwegian University of Science and Technology
Locations (2):
- St Olavs Hospital, Trondheim, Norway
- Lower Umfolozi Rigional War Memorial Hospital, NICU, Empangeni, South Africa

REFERENCES:
- [Result] Kristoffersen L, Malahleha M, Duze Z, Tegnander E, Kapongo N, Stoen R, Follestad T, Eik-Nes SH, Bergseng H. Randomised controlled trial showed that neonates received better pain relief from a higher dose of sucrose during venepuncture. Acta Paediatr. 2018 Dec;107(12):2071-2078. doi: 10.1111/apa.14567. Epub 2018 Oct 2. PMID 30188590